CLINICAL TRIAL: NCT00716547
Title: Multicenter, Randomized, Double-blind, Placebo- and Active-controlled Study of Safety and Efficacy of Two Dosages of Epicutaneously Applied Diractin® (Ketoprofen in Transfersome® Gel) for the Treatment of Osteoarthritis of the Knee
Brief Title: Safety and Efficacy of Two Dosages of Diractin® in Osteoarthritis (OA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IDEA AG (Industry)
Responsible Party: Dr. Claudia Himly / Director of Clinical Operations, IDEA AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL-033-III-03
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ketoprofen; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: ketoprofen in Diractin®
- 2 (Experimental)
  Interventions: Drug: ketoprofen in Diractin®
- 3 (Active Comparator)
  Interventions: Drug: celecoxib
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ketoprofen in Diractin® — 50 mg (b.i.d.)
  Arms: 1
Drug: ketoprofen in Diractin® — 100 mg (b.i.d.)
  Arms: 2
Drug: Placebo — b.i.d.
  Arms: 4
Drug: celecoxib — 100 mg (b.i.d.)
  Arms: 3

SUMMARY:
The purpose of this study is to provide replicated evidence of safety and efficacy of 50 mg and 100 mg ketoprofen in Diractin®.

DETAILED DESCRIPTION:
The study will investigate safety and efficacy of 2 dosages of Diractin®at relieving the signs and symptoms of knee OA, including the primary endpoint of patient assessment of pain.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated
* Age > 45 years
* Class I-III OA of the knee and subject meets American College of Rheumatology (ACR) clinical classification criteria for osteoarthritis of the knee

Exclusion Criteria:

* Skin lesions or dermatological diseases in the treatment area
* Directly or indirectly involved in the conduct and administration of this study
* Received any investigational medicinal product within 30 days prior to Screening Visit or participation in any previous clinical study with Diractin®
* Pregnancy or lactation
* Residents of psychiatric wards, prisons or other state institutions
* Malignancy within the past 2 years
* Depressive disorders requiring treatment with tricyclics, treatment with other antidepressants must be stable for 3 months prior to screening and throughout the study
* Epilepsy
* Schizophrenia
* Neuropathic pain and any other pain condition requiring chronic use of pain medication
* Known hypersensitivity or allergy (including photoallergy) to NSAID´s including ketoprofen, celecoxib, sulfonamides and ingredients used in pharmaceutical products including galactose
* Peripheral arterial disease and/or cerebrovascular disease
* History of stroke or myocardial infarction
* Congestive Heart failure NYHA Class II-IV
* History of pancreatitis or peptic ulcers;
* Inflammatory GI disease (e.g. M. Crohn, colitis ulcerosa)
* Serum creatinine levels > 2.5 milligrams/deciliter (mg/dL)
* ALT or AST levels ≥ 5 times the ULN
* Unable to discontinue analgesic therapy including opioids, NSAID´s, tramadol, muscle relaxants, gabapentin, pregabalin, duloxetine, venlafaxine, capsaicine or other drugs approved or used for the treatment of pain for the duration of the study

Min Age: 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1399 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
pain subscale of the WOMAC | week 12

SECONDARY OUTCOMES:
Patient global assessment of response to therapy | week 12
function subscale of the WOMAC | week 12

CONTACTS AND LOCATIONS:
Overall Officials: IDEA AG Clinical Trial, Study Director — IDEA AG
Locations (4):
- IDEA Investigational Site, Prague, Czechia
- Klaus-Miehlke-Klinik, Wiesbaden, Germany
- NZOZ Nasz Lekarz, Torun, Poland
- Chapel Allerton Hospital, Leeds, United Kingdom

REFERENCES:
- [Derived] Conaghan PG, Dickson J, Bolten W, Cevc G, Rother M. A multicentre, randomized, placebo- and active-controlled trial comparing the efficacy and safety of topical ketoprofen in Transfersome gel (IDEA-033) with ketoprofen-free vehicle (TDT 064) and oral celecoxib for knee pain associated with osteoarthritis. Rheumatology (Oxford). 2013 Jul;52(7):1303-12. doi: 10.1093/rheumatology/ket133. Epub 2013 Mar 28. PMID 23542612